CLINICAL TRIAL: NCT02276456
Title: The Impact of Early Versus Standard Post-Discharge Follow-up on Readmission Rates in Patients Admitted With Myocardial Infarction
Brief Title: The Impact of Early Follow-up on Readmission Rates in AMI Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00046405
Record Dates: First submitted 2014-10-01; First posted 2014-10-28 (Estimated); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- early follow-up (Experimental): Follow-up within 7 days after discharge from hospital after having an MI. This will be the early-follow-up or experimental arm.
  Interventions: Behavioral: Follow-up Appointment- early vs standard
- standard follow-up (No Intervention): Follow-up appointment within 14-18 days after discharge from hospital after having an MI

INTERVENTIONS:
Behavioral: Follow-up Appointment- early vs standard — Patient will undergo early follow-up (within 7 days of discharge) of discharge
  Arms: early follow-up

SUMMARY:
With no prior prospective study to demonstrate the benefit of an early post-discharge follow-up appointment in reducing readmission rates in the post-myocardial infarction (MI patient population, we propose to conduct the first randomized, prospective trial to better elucidate the association between early and standard follow-up on readmission rates. The investigators hypothesize that unlike heart failure or advanced valvular disease patients, the benefit of early outpatient follow-up in reducing readmission of post-MI patients will be less clear. Thus, the investigators primary aim will be to determine the effect of early outpatient follow-up post-discharge on 90 day all-cause readmission rates (exclusive of planned readmissions known at the time of discharge). Secondary aims are to describe 1) causes of readmissions within 90 days, 2) any cardiovascular-related complications and any deaths that occur from discharge through 90 days, 3) 30-day readmission rates and 4) median time to readmission among those readmitted. Finally, the investigators will examine the distribution of demographic, clinical and socioeconomic characteristic according to readmission vs. no readmission. The investigators do not expect to have sufficient endpoints for full predictive modeling, but believe this exploratory work will provide a foundation for future studies. The investigators postulate that the design and methodology of our current study could be used to answer similar questions in other subsets of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute MI (STEMI or NSTEMI) will be recruited from the PAC-CCU service and may have been admitted through the Duke Emergency Department or transferred from a referring hospital. - Clinical events and treatment during the hospitalization (e.g., medical management versus cardiac catheterization, ICU vs. non-ICU care, choice of medications, etc.) will not influence inclusion in the trial and inclusion in the trial will not influence treatment during hospitalization or during follow up, except for the timing of the follow-up appointment.

Exclusion Criteria:

* Patients treated with coronary artery bypass grafting will be excluded for the purposes of this trial to avoid conflicts with usual post-operative management.
* Additionally, patients with features or clinical courses that would preclude the possibility of readmission will be excluded.
* Examples include transition of care goals to comfort care, transition of care to inpatient or outpatient hospice, or the development of complications during the hospitalization that require early follow up appointments (e.g., diagnosis of malignancy).
* Patients discharged to skilled nursing facilities will be eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2014-03; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
hospital readmission | within 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Newby, Principal Investigator — Duke Clinical Research Institute
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States